CLINICAL TRIAL: NCT00783770
Title: Comparison of Monosaccharide Content of Maternal and Umbilical Venous Cord Blood in Term and Preterm Pregnancies
Brief Title: Maternal and Infant Cord Blood Monosaccharide Content
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); University of Arkansas (Other)
Responsible Party: Joanne S. Szabo, M.D., University of Arkansas for Medical Sciences
Other Study IDs: 31247
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Pregnancy
Keywords: Breastfeeding; Infant; Preterm; Nutrition
MeSH Terms: conditions — Breast Feeding; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma will be stored
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 30-33 weeks: mother infant pairs with gestation of 30-33 weeks
- 34-37 weeks: mother infant pairs with gestation of 34-37 weeks
- 38-42 weeks: mother infant pairs with gestation of 38-42 weeks

SUMMARY:
Mother's breast milk provides many benefits to babies with regard to development and improved health. We believe the simple sugars which make up these complex sugars in breast milk and are also found in the brain may be critical to normal brain development in term and preterm infants.

Babies are exposed to these sugars by placental transport during pregnancy and through mother's breast milk after they are born. For the preterm infant, we do not know if breast milk gives enough of these sugars compared to what the baby gets during pregnancy.

A maternal blood sample and blood samples from the baby's umbilical cord will provide us with background information for developing a supplement of special sugars that can be added to infant formulas to provide the amount that the baby usually gets during pregnancy and from breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Healthy mothers with ages ranging from 18 to 35 yrs
* Delivered infants appropriate weight for gestational age (between 10% and 90%)

Exclusion Criteria:

* Maternal history of smoking, alcohol or drug use

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Twenty-four generally healthy mother-infant pairs.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2005-07; Primary Completion 2007-03 (Actual)